CLINICAL TRIAL: NCT00236678
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess Fatigue in Patients With Anemia of Chronic Disease (ACD) Due to Rheumatoid Arthritis Receiving PROCRIT� (Epoetin Alfa)
Brief Title: Randomized, Double-blind, Placebo-controlled Study to Assess Fatigue in Patients With ACD Due to RA Receiving PROCRIT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to slow enrollment, despite protocol amendments to change the entrance criteria.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004624
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-03

CONDITIONS: Anemia; Rheumatoid Arthritis
Keywords: Anemia; Rheumatoid arthritis; Hemoglobin level
MeSH Terms: conditions — Anemia; Arthritis, Rheumatoid | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this research study is to determine fatigue (tiredness) in subjects with chronic Rheumatoid Arthritis with chronic anemia. Fatigue in subjects who get PROCRIT will be compared to fatigue in subjects who get placebo (a medically inactive substance). The study will also evaluate hemoglobin levels (oxygen-carrying protein in red blood cells), safety, anemia related health concerns, vitality, arthritis related function and work productivity.

DETAILED DESCRIPTION:
PROCRIT is not approved for the treatment of anemia of chronic disease in rheumatoid arthritis patients.

Approximately 270 subjects will be participating in this trial, at approximately 25 centers in the United States. Patients will be eligible to participate in this study if hemoglobin (Hb) is <=11.0 g/dL. The hypothesis is that PROCRIT improves fatigue scores in rheumatoid arthritis patients with anemia of chronic disease. If a patient chooses to participate, he/she will be randomized to receive either PROCRIT or placebo on a weekly basis starting at 20,000 units per injection (up to a maximum of 40,000 units).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have rheumatoid arthritis with chronic anemia. Patients must have signed an informed consent
* women must be postmenopausal for at least one year, surgically sterile, or practicing an effective method of birth control, or have a negative serum pregnancy test
* women must not be breast feeding during this study period.

Exclusion Criteria:

* Uncontrolled hypertension
* elective surgery, including joint replacement, anticipated to require transfusion during the extension study period
* thromboembolic event during the double-blind study including acute myocardial infarction, cerebrovascular accident and/or transient ischemic attack
* deep vein thrombosis and/or pulmonary embolism
* uncontrolled psychiatric disease
* planning to be enrolled in any other clinical trial during the course of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-07; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To assess changes in fatigue in patients at least 18 years old with chronic rheumatoid arthritis (RA) and chronic anemia (Hb < 11.0 g/dL) due to ACD receiving weekly s.c. doses of PROCRIT versus placebo.

SECONDARY OUTCOMES:
Hb response; changes in anemia associated health concerns; changes in vitality; changes in arthritis related function

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Randomized, Double-blind, Placebo-controlled Study to Assess Fatigue in Patients with Anemia of Chronic Disease (ACD) Due to Rheumatoid Arthritis Receiving PROCRIT (Epoetin alfa) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=609&filename=CR004624_CSR.pdf